CLINICAL TRIAL: NCT02854176
Title: Somatosensory Electrical Stimulation to Improve Motor Control in Patients Suffering From Knee Osteoarthritis
Brief Title: Somatosensory Stimulation in Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Menno Veldman (Other)
Collaborators: Schulthess Klinik (Other)
Responsible Party: Sponsor-Investigator, Menno Veldman, MSc, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: Somatosensory stimulation
Record Dates: First submitted 2016-07-26; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Somatosensory electrical stimulation (Experimental)
  Interventions: Procedure: Somatosensory electrical stimulation
- Control (Sham Comparator)
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Somatosensory electrical stimulation
  Arms: Somatosensory electrical stimulation
Procedure: Control
  Arms: Control

SUMMARY:
Worldwide, 9.6% of men and 18% of women aged over 60 years suffer from osteoarthritis (OA), most of which involve the knee. Within the OA patient population, 80% of the OA patients have limitations of movement, and 25% cannot perform the majority of their daily activities (WHO). Some of these symptoms contribute to arthrogenic muscle inhibition (AMI), a reflexive decrease in motor output to the muscles surrounding the affected joint.

AMI is characterized by abnormal afferent information transmitted to the central nervous system, resulting in altered afferent feedback to the quadriceps motoneurons (MN) which in turn results in reduced excitability of that particular pool. The altered afferent input is suggested to stem from stimulation of mechanoreceptors, via joint effusion or excessive movements, nociceptors as a response to pain, or loss of joint receptors (Palmieri-Smith et al., 2009). Although the evidence concerning the role of the central nervous system is scarce, pre- and postsynaptic spinal mechanisms directly affecting alpha-MNs seem affected. Dysfunction of γ-loops also seems to be involved (Konishi et al., 2002). These mechanisms together result in AMI that manifests through aberrations in voluntary quadriceps torque, force control, and reflex excitability often measured by the H-reflex (Hopkins et al., 2000).

Besides the evident role of motor efferents, sensory afferents also influence motor control (Gentilucci et al., 1997) and poor proprioceptive function is predictive of poor chair-stand performance (Sharma et al., 2003). Reduction of the sensory deficits could potentially increase motor function in knee OA. The present study aims to evaluate whether low-intensity peripheral electrical nerve stimulation, a form of increasing afferent input, could potentially improve OA patients' motor function. The most limiting factor in OA patients, however, is pain, experienced at rest and during movement. Although previous paradigms used high-frequency stimulation and the lack of physiological explanations concerning pain reductions after peripheral electrical nerve stimulation, it is possible that reductions in experienced pain are mediated by reduced analgesia, i.e., decreased excitability of nociceptive neurons.

DETAILED DESCRIPTION:
Worldwide, 9.6% of men and 18% of women aged over 60 years suffer from osteoarthritis (OA), most of which involve the knee. Within the OA patient population, 80% of the OA patients have limitations of movement, and 25% cannot perform the majority of their daily activities (WHO). OA is a progressive articular cartilage disorder involving motor and sensory dysfunctions, including a decreased range of motion, muscle weakness, impaired proprioception, and pain. Some of these symptoms contribute to arthrogenic muscle inhibition (AMI), a reflexive decrease in motor output to the muscles surrounding the affected joint that is most likely mediated by GABAergic inhibitory mechanisms.

AMI is characterized by abnormal afferent information transmitted to the central nervous system, resulting in altered afferent feedback to the quadriceps motoneurons (MN) which in turn results in reduced excitability of that particular pool. The altered afferent input is suggested to stem from stimulation of mechanoreceptors, via joint effusion or excessive movements, nociceptors as a response to pain, or loss of joint receptors. Although the evidence concerning the role of the central nervous system is scarce, pre- and postsynaptic spinal mechanisms directly affecting alpha-MNs seem affected. Dysfunction of γ-loops also seems to be involved. These mechanisms together result in AMI that manifests through aberrations in voluntary quadriceps torque, force control, and reflex excitability often measured by the H-reflex.

Motor dysfunction thus is an important limiting factor for OA patients and involves motor and sensory factors. Besides the evident role of motor efferents, sensory afferents also influence motor control and poor proprioceptive function is predictive of poor chair-stand performance. Reduction of the sensory deficits could potentially increase motor function in knee OA. The present study aims to evaluate whether low-intensity peripheral electrical nerve stimulation, a form of increasing afferent input, could potentially improve OA patients' motor function. The most limiting factor in OA patients, however, is pain, experienced at rest and during movement. High-frequencies stimulation paradigms are normally used to reduce pain, but 40-50 minutes of low-frequency electrical stimulation (4 Hz, < MT intensity) can also be effective in reducing pain at rest, pain during movement, and pain sensitivity, although a recent systematic review questions consistency of these effects considering the limited evidence. Although, to the best of our knowledge, there is no clear physiological explanation concerning pain reductions after peripheral electrical nerve stimulation, it is possible that reductions in experienced pain are mediated by reduced analgesia, i.e., decreased excitability of nociceptive neurons.

Electrical stimulation of peripheral nerves and muscles has been applied in various forms to modulate muscle strength, motor skill, spinal- and cortical excitability. Neuromuscular electrical stimulation (NMES) evoked forces can generate torques up to 112% of maximal voluntary contraction force and increases with increasing stimulation frequency up to 70-80 Hz.

Whereas NMES is primarily focused on increasing muscle strength, low-intensity somatosensory electrical stimulation (SES) has been used to increase motor skill acquisition in neurologic patients and healthy participants. SES excites group Ia, Ib, and II afferents, as well as secondary muscle afferent fibers. SES increases motor performance the most when applied to a peripheral nerve at high sensory intensities (2-3 times perceptual threshold) at 10 Hz (SES applied in 1 Hz trains consisting of 5 pulses at 10 Hz). High-frequency transcutaneous electrical nerve stimulation (TENS) and sensorimotor training can both repositioning error reflecting impaired knee proprioception in patients with knee OA. Both TENS and SES thus excite afferent fibers involved in knee proprioception. Impaired knee proprioception has been associated with impaired ability to accurately and steadily control force and impaired eccentric strength. In contrast with NMES, in which induced increases in muscle force most likely involve changes in metabolism, hypertrophy, and possibly spinal mechanisms, and TENS, where large diameter primary afferents are pivotal in pain reductions, SES targets sensory pathways, both cutaneous and proprioceptive, which seem an appropriate target to reduce sensory deficits involved in OA.

SES can improve stroke patients' motor function but whether such improvements can occur in patients with knee AO is unknown. Excitation of primary afferents by SES could serve as a physiological basis for the hypothesis that SES positively influences the afferent input to α-MN of the quadriceps muscles surrounding the dysfunctional joint and reduce pain. The increased afferent input by SES, as shown previously in healthy participants and stroke patients, is expected to increase motor control, measured by an increase in tracking performance in the dysfunctional knee joint. As a task variant to visuomotor tracking, force steadiness and accuracy are expected to increase after SES because these measures are associated with proprioception, an outcome SES is known to improve through excitation of muscle afferents. If this expectation is correct, SES could then be used in future studies and rehabilitation protocols as a primer to potentiate the effects of NMES and other exercise therapies designed to improve quadriceps strength and power. Second, if SES reduces pain and increases motor control, SES can possibly postpone surgery and can serve as an adjuvant for patients for patients who are unsuitable for or resist a total knee replacement to improve activities of daily and therefore quality of life.

Therefore, the present study will examine the acute and delayed effects of 60 minutes of SES (five pulses in 1 Hz trains at 10 Hz at motor threshold intensity) of the femoral nerve in patients suffering from knee OA. Figure 1 depicts a schematic overview of the proposed study design. As an initial step, a pilot experiment in 5-6 healthy individuals should reveal whether there are some effects or trends observed after 30 minutes of SES, a duration probably would be more optimal at 60 minutes considering the 120 minutes standard used for improving neurological patients' hand function. The primary outcomes of the study is motor coordination evaluated using target tracking based on knee position and not based on quadriceps force, because position vs. force is less affected by the influences of pain and therefore more suitable in the current context. Secondary outcomes are motor control and proprioception reflected by increased force steadiness and accuracy, maximal voluntary strength and daily physical function. The investigators hypothesize based on previous data that afferent input induced by SES reduces abnormalities in sensory input as a result of OA, and therefore increases motor control.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years.
* Unilateral symptomatic KOA.
* Patient in waitlist at the Schulthess Clinic for knee arthroplasty.
* Patient has mild to average pain levels
* Living place: Canton of Zurich or neighbouring Cantons.
* Signed written informed consent.

Exclusion Criteria:

* Symptomatic OA in lower extremity joints other than the knee.
* Bilateral symptomatic KOA.
* Usage of walking aids.
* Surgery to the lower limbs in the prior 12 months.
* BMI >35 kg/m2.
* Disorders that affect visuomotor function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Mean absolute deviation from a preprogrammed template during target tracking with the injured knee | Change from before to after 60 minutes of somatosensory electrical stimulation applied to the femoral nerve

SECONDARY OUTCOMES:
Quadriceps force accuracy and steadiness of the injured leg during isometric force at 50 and 100 Newton | Change from before to after 60 minutes of somatosensory electrical stimulation applied to the femoral nerve

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celnik P, Hummel F, Harris-Love M, Wolk R, Cohen LG. Somatosensory stimulation enhances the effects of training functional hand tasks in patients with chronic stroke. Arch Phys Med Rehabil. 2007 Nov;88(11):1369-76. doi: 10.1016/j.apmr.2007.08.001. PMID 17964875
- [Background] Courtney CA, O'Hearn MA, Hornby TG. Neuromuscular function in painful knee osteoarthritis. Curr Pain Headache Rep. 2012 Dec;16(6):518-24. doi: 10.1007/s11916-012-0299-2. PMID 23054978
- [Background] Gentilucci M, Toni I, Daprati E, Gangitano M. Tactile input of the hand and the control of reaching to grasp movements. Exp Brain Res. 1997 Mar;114(1):130-7. doi: 10.1007/pl00005612. PMID 9125458
- [Background] Herzig D, Maffiuletti NA, Eser P. The Application of Neuromuscular Electrical Stimulation Training in Various Non-neurologic Patient Populations: A Narrative Review. PM R. 2015 Nov;7(11):1167-1178. doi: 10.1016/j.pmrj.2015.03.022. Epub 2015 Mar 31. PMID 25839763
- [Background] Hopkins JT, Ingersoll CD, Edwards JE, Cordova ML. Changes in soleus motoneuron pool excitability after artificial knee joint effusion. Arch Phys Med Rehabil. 2000 Sep;81(9):1199-203. doi: 10.1053/apmr.2000.6298. PMID 10987162
- [Background] Hortobagyi T, Garry J, Holbert D, Devita P. Aberrations in the control of quadriceps muscle force in patients with knee osteoarthritis. Arthritis Rheum. 2004 Aug 15;51(4):562-9. doi: 10.1002/art.20545. PMID 15334428
- [Background] Hortobagyi T, Scott K, Lambert J, Hamilton G, Tracy J. Cross-education of muscle strength is greater with stimulated than voluntary contractions. Motor Control. 1999 Apr;3(2):205-19. doi: 10.1123/mcj.3.2.205. PMID 10198150
- [Background] Kaelin-Lang A. Enhancing rehabilitation of motor deficits with peripheral nerve stimulation. NeuroRehabilitation. 2008;23(1):89-93. PMID 18356592
- [Background] Kaelin-Lang A, Luft AR, Sawaki L, Burstein AH, Sohn YH, Cohen LG. Modulation of human corticomotor excitability by somatosensory input. J Physiol. 2002 Apr 15;540(Pt 2):623-33. doi: 10.1113/jphysiol.2001.012801. PMID 11956348
- [Background] Konishi Y, Fukubayashi T, Takeshita D. Mechanism of quadriceps femoris muscle weakness in patients with anterior cruciate ligament reconstruction. Scand J Med Sci Sports. 2002 Dec;12(6):371-5. doi: 10.1034/j.1600-0838.2002.01293.x. PMID 12453165
- [Background] Maffiuletti NA, Bizzini M, Schatt S, Munzinger U. A multi-joint lower-limb tracking-trajectory test for the assessment of motor coordination. Neurosci Lett. 2005 Aug 12-19;384(1-2):106-11. doi: 10.1016/j.neulet.2005.04.064. PMID 15885904
- [Background] Palmieri-Smith RM, Thomas AC. A neuromuscular mechanism of posttraumatic osteoarthritis associated with ACL injury. Exerc Sport Sci Rev. 2009 Jul;37(3):147-53. doi: 10.1097/JES.0b013e3181aa6669. PMID 19550206
- [Background] Poortvliet PC, Tucker KJ, Finnigan S, Scott D, Sowman P, Hodges PW. Cortical activity differs between position- and force-control knee extension tasks. Exp Brain Res. 2015 Dec;233(12):3447-57. doi: 10.1007/s00221-015-4404-8. Epub 2015 Aug 21. PMID 26292962
- [Background] Radhakrishnan R, Sluka KA. Deep tissue afferents, but not cutaneous afferents, mediate transcutaneous electrical nerve stimulation-Induced antihyperalgesia. J Pain. 2005 Oct;6(10):673-80. doi: 10.1016/j.jpain.2005.06.001. PMID 16202960
- [Background] Roos EM, Klassbo M, Lohmander LS. WOMAC osteoarthritis index. Reliability, validity, and responsiveness in patients with arthroscopically assessed osteoarthritis. Western Ontario and MacMaster Universities. Scand J Rheumatol. 1999;28(4):210-5. doi: 10.1080/03009749950155562. PMID 10503556
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417
- [Background] Sharma L, Cahue S, Song J, Hayes K, Pai YC, Dunlop D. Physical functioning over three years in knee osteoarthritis: role of psychosocial, local mechanical, and neuromuscular factors. Arthritis Rheum. 2003 Dec;48(12):3359-70. doi: 10.1002/art.11420. PMID 14673987
- [Background] Shirazi ZR, Shafaee R, Abbasi L. The effects of transcutaneous electrical nerve stimulation on joint position sense in patients with knee joint osteoarthritis. Physiother Theory Pract. 2014 Oct;30(7):495-9. doi: 10.3109/09593985.2014.903547. Epub 2014 Apr 3. PMID 24697730
- [Background] Smith JW, Marcus RL, Peters CL, Pelt CE, Tracy BL, LaStayo PC. Muscle force steadiness in older adults before and after total knee arthroplasty. J Arthroplasty. 2014 Jun;29(6):1143-8. doi: 10.1016/j.arth.2013.11.023. Epub 2013 Dec 2. PMID 24405624
- [Background] Tsauo JY, Cheng PF, Yang RS. The effects of sensorimotor training on knee proprioception and function for patients with knee osteoarthritis: a preliminary report. Clin Rehabil. 2008 May;22(5):448-57. doi: 10.1177/0269215507084597. PMID 18441041
- [Background] Vance CG, Rakel BA, Blodgett NP, DeSantana JM, Amendola A, Zimmerman MB, Walsh DM, Sluka KA. Effects of transcutaneous electrical nerve stimulation on pain, pain sensitivity, and function in people with knee osteoarthritis: a randomized controlled trial. Phys Ther. 2012 Jul;92(7):898-910. doi: 10.2522/ptj.20110183. Epub 2012 Mar 30. PMID 22466027
- [Background] Veldman MP, Zijdewind I, Solnik S, Maffiuletti NA, Berghuis KM, Javet M, Negyesi J, Hortobagyi T. Direct and crossed effects of somatosensory electrical stimulation on motor learning and neuronal plasticity in humans. Eur J Appl Physiol. 2015 Dec;115(12):2505-19. doi: 10.1007/s00421-015-3248-z. Epub 2015 Sep 3. PMID 26335625
- [Background] Veldman MP, Zijdewind I, Maffiuletti NA, Hortobagyi T. Motor Skill Acquisition and Retention after Somatosensory Electrical Stimulation in Healthy Humans. Front Hum Neurosci. 2016 Mar 16;10:115. doi: 10.3389/fnhum.2016.00115. eCollection 2016. PMID 27014043
- [Background] Wu CW, Seo HJ, Cohen LG. Influence of electric somatosensory stimulation on paretic-hand function in chronic stroke. Arch Phys Med Rehabil. 2006 Mar;87(3):351-7. doi: 10.1016/j.apmr.2005.11.019. PMID 16500168